CLINICAL TRIAL: NCT06733246
Title: Evaluation of the Safey & Performance of the Ceretrieve Device Designed for Thrombus Removal in Intracranial Arteries Using an Aspiration Technique in Patients Suffering an Acute Ischemic Stroke (AIS)
Brief Title: Safety and Efficacy Evaluation of the Ceretrieve Device in the Treatment of AIS Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ceretrieve Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA 304
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Thrombectomy; Aspiration; Neuro-thrombectomy catheter; stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ceretrieve treatment arm - patient will be treated with the Ceretrieve device - aspiration approach (Experimental): This is the only study arm. All patients found to be eligible will be treated with the Ceretrieve device.
  Interventions: Device: Aspiration 0

INTERVENTIONS:
Device: Aspiration 0 — Ceretrieve is a neuro-thrombectomy aspiration catheter deigned for clot removal in AIS patients.

SUMMARY:
The main objective of this clinical trial is to evaluate of the safety & efficacy of the Ceretrieve device within 24 hours post thrombectomy procedure. This means to assess that the use with the Ceretrieve neuro-thrombectomy device that is designed to treat acute ischemic stroke patients raises no safety concerns and that it is found to be effective when it is used according to its intended purpose, which is revascularization of patients with acute ischemic stroke secondary to intracranial large vessel occlusive disease (involving the internal carotid artery, middle cerebral artery- M1 and M2 segments, basilar, and vertebral arteries).

The study researchers will compare the efficacy and safety results of this study to data derived from the literature of FDA approved neuro-thrombectomy devices. The study hypothesis is that The Ceretrieve device would achieve successful reperfusion performance shall be similar to the safety & performance derived from the literature.

The primary outcomes that will be measures are:

Performance:

Successful reperfusion, defined as core laboratory-adjudicated modified Thrombolysis in Cerebral Ischemia (mTICI) score 2b-3 within three passes of the Ceretrieve system without any rescue.

Safety:

Symptomatic intra-cranial hemorrhage within 24 (18-36) hours of the study procedure.

Patients who will participate in this study will be followed for a time period of 3 months. After discharge from the medical center, they will be asked to arrive to a one visit at the clinic for safety data collection and evaluation.

DETAILED DESCRIPTION:
This study is designed as a prospective, multi-center, open-label, single-arm study.

Patient will be required to undergo screening evaluation to confirm he/she meet the eligibility study criteria and are suitable to be a study participant.

The study patient population is comprised of adult subjects 18 years old and above, suffering from acute ischemic stroke, with a new moderate-to-severe neurologic deficits, angiographically confirmed occlusion in the intracranial internal carotid, middle cerebral (M1 or M2 segment), basilar, or vertebral artery, and can undergo endovascular therapy (at least one Ceretrieve deployment in the target artery), within 24 hours of symptoms on set.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age
2. Clinical signs consistent with acute ischemic stroke
3. Subject is able to be treated within 24 hours of stroke symptom onset.
4. Pre-stroke modified Rankin Score of 0 or 1
5. NIHSS > 6 at the time of screening
6. If intravenous thrombolysis (IVT) is indicated, initiation of IVT should be administered as soon as possible and no later than 4.5 hours of onset of stroke symptoms (onset time is defined as the last time when the patient was witnessed to be at baseline neurologic status), with investigator verification that the subject has received/is receiving the correct IVT dose for the estimated weight.
7. Intracranial occlusion defined as Modified Thrombolysis in Cerebral Infarction (mTICI) 0-1 flow confirmed by angiography that is accessible to the mechanical thrombectomy device in the following locations:

1. Intracranial internal carotid artery 2. M1 and/or M2 segment of the MCA 3. Vertebral artery 4. Basilar artery Note: M1 segment of the MCA is defined as the arterial trunk from its origin at the ICA to the first bifurcation or trifurcation into major branches neglecting the small temporo-polar branch.

8. A valid completed informed consent in accordance with the local ethics committee regulations.

Exclusion Criteria:

1. Female who is pregnant or lactating or has a positive pregnancy test at time of admission.
2. Rapid neurological improvement prior to study enrolment suggesting resolution of signs/symptoms of stroke
3. Known serious sensitivity to radiographic contrast agents
4. Known sensitivity to nickel, titanium metals, or their alloys
5. Subjects already enrolled in other investigational studies that would interfere with study endpoints
6. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency. (A subject without history or suspicion of coagulopathy does not require INR or prothrombin time lab results to be available prior to enrolment.)
7. Life expectancy of less than 90 days
8. Clinical presentation suggests a subarachnoid hemorrhage, even if the initial CT or MRI scan is normal.
9. Suspicion of aortic dissection
10. Subject with a comorbid disease or condition that would confound the neurological and functional evaluations or compromise survival or ability to complete follow-up assessments.
11. Known to currently use or abuses alcohol (defined as regular or daily consumption of more than four alcoholic drinks per day).
12. Known arterial condition (e.g., proximal vessel stenosis or pre-existing stent) that would prevent the device from reaching the target vessel and/or preclude safe recovery of the device
13. Subject who requires balloon angioplasty or stenting of the carotid artery at the time of the index procedure
14. Angiographic evidence of carotid dissection
15. Imaging exclusion criteria:

    * CT or MRI evidence of hemorrhage on presentation
    * CT or MRI evidence of mass effect or intra-cranial tumor (except small meningioma)
    * CT or MRI evidence of cerebral vasculitis
    * CT or MRI-DWI showing ASPECTS 0-5 (or pc-ASPECTS 0-6 in the posterior circulation). Alternatively, if automated core volume assessment software is used, MRI-DWI or CTP core > 70cc.
    * CT/MRI shows evidence of carotid dissection or complete cervical carotid occlusion requiring a stent
    * Any imaging evidence that suggests, in the opinion of the investigator, that the subject is not appropriate for mechanical thrombectomy intervention while utilizing an aspiration approach (e.g. inability to navigate to the target lesion, moderate/large infarct with poor collateral circulation, etc.).
16. Occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation) as confirmed by angiography, or clinical evidence of bilateral strokes or strokes in multiple territories.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy | intra-procedural
  Successful reperfusion, defined as core laboratory-adjudicated modified Thrombolysis in Cerebral Ischemia (mTICI) score 2b-3 within three passes of the Ceretrieve system without any rescue.
Safety | 24 (18-36) hours post procedure
  Symptomatic Intra-cranial hemorrhage within 24 (18-36) hours post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Heidelberg University Hospital, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No
All data in the study will undergo pseudo-anonymization process and there will be no identifiable details in the data collected on all study patients.
  In this study, all endpoints are aimed at assessing/analyzing events' rates to be compared against the applicable historical data, and not the review of individual cases data.

REFERENCES:
- [Background] Turk AS 3rd, Siddiqui A, Fifi JT, De Leacy RA, Fiorella DJ, Gu E, Levy EI, Snyder KV, Hanel RA, Aghaebrahim A, Woodward BK, Hixson HR, Chaudry MI, Spiotta AM, Rai AT, Frei D, Almandoz JED, Kelly M, Arthur A, Baxter B, English J, Linfante I, Fargen KM, Mocco J. Aspiration thrombectomy versus stent retriever thrombectomy as first-line approach for large vessel occlusion (COMPASS): a multicentre, randomised, open label, blinded outcome, non-inferiority trial. Lancet. 2019 Mar 9;393(10175):998-1008. doi: 10.1016/S0140-6736(19)30297-1. PMID 30860055
- [Background] Guo X, Xiong Y, Huang X, Pan Z, Kang X, Chen C, Zhou J, Wang C, Lin S, Hu W, Wang L, Zheng F. Aspiration versus stent retriever for posterior circulation stroke: A meta-analysis. CNS Neurosci Ther. 2023 Feb;29(2):525-537. doi: 10.1111/cns.14045. Epub 2022 Dec 13. PMID 36513959
- [Background] Jolugbo P, Ariens RAS. Thrombus Composition and Efficacy of Thrombolysis and Thrombectomy in Acute Ischemic Stroke. Stroke. 2021 Mar;52(3):1131-1142. doi: 10.1161/STROKEAHA.120.032810. Epub 2021 Feb 10. PMID 33563020
- [Background] Pilgram-Pastor SM, Piechowiak EI, Dobrocky T, Kaesmacher J, Den Hollander J, Gralla J, Mordasini P. Stroke thrombectomy complication management. J Neurointerv Surg. 2021 Oct;13(10):912-917. doi: 10.1136/neurintsurg-2021-017349. Epub 2021 Jun 22. PMID 34158401
- [Background] Baek JH, Kim BM, Kang DH, Heo JH, Nam HS, Kim YD, Hwang YH, Kim YW, Kim YS, Kim DJ, Kwak HS, Roh HG, Lee YJ, Kim SH, Baik SK, Jeon P, Yoo J, Suh SH, Kim B, Kim JW, Suh S, Jeon HJ. Balloon Guide Catheter Is Beneficial in Endovascular Treatment Regardless of Mechanical Recanalization Modality. Stroke. 2019 Jun;50(6):1490-1496. doi: 10.1161/STROKEAHA.118.024723. Epub 2019 May 2. PMID 31043149
- [Background] Kim YW, Hwang YH, Kim YS, Kang DH. Frontline contact aspiration thrombectomy using SOFIA catheter for acute ischemic stroke: period-to-period comparison with Penumbra catheter. Acta Neurochir (Wien). 2019 Jun;161(6):1197-1204. doi: 10.1007/s00701-019-03914-4. Epub 2019 Apr 29. PMID 31037498
- [Background] Fanous AA, Siddiqui AH. Mechanical thrombectomy: Stent retrievers vs. aspiration catheters. Cor Vasa. 2016;58(2):e193-e203. doi:10.1016/j.crvasa.2016.01.004
- [Background] Munich SA, Vakharia K, Levy EI. Overview of Mechanical Thrombectomy Techniques. Neurosurgery. 2019 Jul 1;85(suppl_1):S60-S67. doi: 10.1093/neuros/nyz071. PMID 31197338
- [Background] Huang JC, Bhaskar SMM. Clot Morphology in Acute Ischemic Stroke Decision Making. Int J Mol Sci. 2022 Oct 15;23(20):12373. doi: 10.3390/ijms232012373. PMID 36293230
- [Background] Zaidat OO, Castonguay AC, Linfante I, Gupta R, Martin CO, Holloway WE, Mueller-Kronast N, English JD, Dabus G, Malisch TW, Marden FA, Bozorgchami H, Xavier A, Rai AT, Froehler MT, Badruddin A, Nguyen TN, Taqi MA, Abraham MG, Yoo AJ, Janardhan V, Shaltoni H, Novakovic R, Abou-Chebl A, Chen PR, Britz GW, Sun CJ, Bansal V, Kaushal R, Nanda A, Nogueira RG. First Pass Effect: A New Measure for Stroke Thrombectomy Devices. Stroke. 2018 Mar;49(3):660-666. doi: 10.1161/STROKEAHA.117.020315. Epub 2018 Feb 19. PMID 29459390
- [Background] Patil S, Darcourt J, Messina P, Bozsak F, Cognard C, Doyle K. Characterising acute ischaemic stroke thrombi: insights from histology, imaging and emerging impedance-based technologies. Stroke Vasc Neurol. 2022 Aug;7(4):353-363. doi: 10.1136/svn-2021-001038. Epub 2022 Mar 3. PMID 35241632
- [Background] Haupt M, Gerner ST, Bahr M, Doeppner TR. Neuroprotective Strategies for Ischemic Stroke-Future Perspectives. Int J Mol Sci. 2023 Feb 22;24(5):4334. doi: 10.3390/ijms24054334. PMID 36901765
- [Background] Primiani CT, Vicente AC, Brannick MT, Turk AS, Mocco J, Levy EI, Siddiqui AH, Mokin M. Direct Aspiration versus Stent Retriever Thrombectomy for Acute Stroke: A Systematic Review and Meta-Analysis in 9127 Patients. J Stroke Cerebrovasc Dis. 2019 May;28(5):1329-1337. doi: 10.1016/j.jstrokecerebrovasdis.2019.01.034. Epub 2019 Feb 14. PMID 30772159
- [Background] Wahlgren N, Ahmed N, Davalos A, Ford GA, Grond M, Hacke W, Hennerici MG, Kaste M, Kuelkens S, Larrue V, Lees KR, Roine RO, Soinne L, Toni D, Vanhooren G; SITS-MOST investigators. Thrombolysis with alteplase for acute ischaemic stroke in the Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST): an observational study. Lancet. 2007 Jan 27;369(9558):275-82. doi: 10.1016/S0140-6736(07)60149-4. PMID 17258667